CLINICAL TRIAL: NCT05955469
Title: Comparison of Speech Understanding Between a Tonotopy-based Bimodal Fitting and a Default Bimodal Fitting in Newly Cochlear-implanted Patients: a Double-blind Randomized Crossover Study.
Brief Title: Comparison in New Cochlear Implanted Subjects of a Tonotopy-based Bimodal Fitting and a Conventional Fitting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MEDEL_COTONBIM_StEtienne_study
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Sensorineural Hearing Loss, Bilateral; Bilateral Hearing Loss
Keywords: Cochlear implant; Bimodal fitting; Anatomy-based fitting
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral | interventions — Cochlear Implants

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
  Two arms A and B:
  Arm A: Bimodal patient's fitting with default fitting (FS4) --> 6 weeks use --> tests and bimodal patient's fitting with tonotopy-based fitting (TFS4) --> 6 weeks use --> tests; Arm B: Bimodal patient's fitting with TFS4 --> 6 weeks use --> tests and bimodal patient's fitting with FS4 --> 6 weeks use --> tests
Who Masked: Participant, Investigator
Masking Description: Double blind study: The patient and the Investigator don't know the fitting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FS4 then TFS4 (Active Comparator): Cochlear Implant with FS4 first during 6 weeks then with TFS4 during 6 weeks
  Interventions: Device: FS4 then TFS4 (cochlear implant)
- TFS4 then FS4 (Active Comparator): Cochlear Implant with TFS4 first during 6 weeks then with FS4 during 6 weeks
  Interventions: Device: TFS4 then FS4 (cochlear implant)

INTERVENTIONS:
Device: FS4 then TFS4 (cochlear implant) — Cochlear implant with default fitting then with tonotopy-based fitting
  Arms: FS4 then TFS4
Device: TFS4 then FS4 (cochlear implant) — Cochlear implant with tonotopy-based fitting then with default fitting
  Arms: TFS4 then FS4

SUMMARY:
Main objective:

For a bimodal fitting (hearing aid (HA) + cochlear implant (CI)): Comparison of a tonotopy based fitting strategy (TFS4) to a default fitting strategy (FS4) for the speech recognition in noise.

Secondary objectives:

Comparison of TFS4 to FS4 for speech recognition in quiet. Comparison of TFS4 to FS4 for the auditory skills experienced by the subject.

DETAILED DESCRIPTION:
Introduction:

Cochlear implantation allows the rehabilitation of profound bilateral deafness, restoring speech perception and verbal communication when the traditional hearing aid no longer provides satisfactory hearing gain. A cochlear implant includes an electrode array and its functioning is based on the principle of cochlear tonotopy: Each electrode encodes a frequency spectrum according to its position in the cochlea (high frequencies are assigned to the basal electrodes and low frequencies to the apical electrodes). The cochlear implant thus breaks down the frequency spectrum into a number of frequency bands via bandpass filters corresponding to the number of electrodes in the implant. During the fitting these bands can be modified by the audiologist.

Bimodal hearing refers to the use of a CI in one ear with a HA on the contralateral side. This association allows for adults and children a better perception of speech in quiet and in noise, a better perception of music, hearing comfort, better sound quality, better localization of sound and, consequently, a better quality of life compared to unilateral CI alone. However, there is great variability in the integration process; while some bimodal users show substantial benefits, others receive little or no benefit.

This variability could be due to the mismatch of frequencies (tonotopic shift) between the CI and the contralateral HA.

Recently MED-EL has developed an "anatomy-based fitting" (ABF) strategy based on the tonotopy that allows, from a postoperative scanner, to calculate the theoretical characteristic frequency of neurons stimulated by each electrode contact and to transmit this information to the fitting software of the CI.

This strategy (TFS4) could therefore allow a better integration of information in bimodal hearing and in particular improve the speech recognition in noise compared to a default strategy (FS4).

Main objective:

For a bimodal fitting (hearing aid (HA) + cochlear implant (CI)): Comparison of a tonotopy based fitting strategy (TFS4) to a default fitting strategy (FS4) for the speech recognition in noise.

Secondary objectives:

Comparison of TFS4 to FS4 for speech recognition in quiet. Comparison of TFS4 to FS4 for the auditory skills experienced by the subject.

Plan of the study:

It is a prospective open monocentric randomized crossover study: Measures will be done on the patient at 6 weeks and 12 weeks post-activation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>= 18 years old) speaking French
* Patient who fulfils the criteria for cochlear implantation

Exclusion Criteria:

* retro-cochlear pathology: auditory neuropathy, vestibular schwannoma
* patient with residual hearing < 70 dB hearing level (HL) at 500 Hz and 1000 Hz on the contralateral ear

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Speech recognition in noise | at 6 weeks post-activation
  The speech recognition in noise is evaluated with the French Matrix test (Framatrix) [S. Jansen et al. Comparison of three types of French speech-in-noise tests: a multi-center study. Int J Audiol, 51 (3) (2012), pp. 164-173].
Speech recognition in noise | at 12 weeks post-activation
  The speech recognition in noise is evaluated with the French Matrix test (Framatrix) [S. Jansen et al. Comparison of three types of French speech-in-noise tests: a multi-center study. Int J Audiol, 51 (3) (2012), pp. 164-173].

SECONDARY OUTCOMES:
Speech recognition in quiet | at 6 weeks post-activation
  Cochlear list of Lafon: list of 51 phonems (17 words). Speech recognition score on 50.
Speech recognition in quiet | at 12 weeks post-activation
  Cochlear list of Lafon: list of 51 phonems (17 words). Speech recognition score on 50.
Auditory skills experienced by the patient | at 6 weeks post-activation
  Auditory skills experienced by the patient are evaluated with the short form of the French version of the speech spatial qualities scale (SSQ) with of 15 questions describing various real-world auditory situations [Moulin et al. Ear & Hearing 2019;40;938-950].
Auditory skills experienced by the patient | at 12 weeks post-activation
  Auditory skills experienced by the patient are evaluated with the short form of the French version of the speech spatial qualities scale (SSQ) with of 15 questions describing various real-world auditory situations [Moulin et al. Ear & Hearing 2019;40;938-950].

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Karkas, Pr, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No